CLINICAL TRIAL: NCT05695196
Title: Feasibility and Safety Study of Parent-to-Child Nasal Microbiota Transplant to Promote Colonization Resistance to Staphylococcus Aureus
Brief Title: Feasibility and Safety Study of Parent-to-Child Nasal Microbiota Transplant
Acronym: ParentsTREAT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00361302; R21AI179644 (NIH)
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Staphylococcus Aureus; Microbial Colonization; Neonatal Infection
Keywords: microbiome
MeSH Terms: conditions — Staphylococcal Infections; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- direct NMT (Experimental): swab parent nares then insert swab directly into neonate nares
  Interventions: Biological: nasal microbiota transplant (NMT)
- indirect NMT (Experimental): swab parent nares, inoculate swab into saline, instill liquid into neonate nares
  Interventions: Biological: nasal microbiota transplant (NMT)
- placebo (Placebo Comparator): instill sterile saline into neonate nares
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: nasal microbiota transplant (NMT) — nasal microbiota transplant
  Arms: direct NMT; indirect NMT
Biological: Placebo — Placebo sterile saline
  Arms: placebo

SUMMARY:
This feasibility and safety pilot study looks to determine whether transferring a parents healthy, diverse nasal microbiota to the participant's infant(s) will create a healthy, diverse neonatal nasal microbiome.

DETAILED DESCRIPTION:
The parent-to-child NMT study is a pilot study to test the feasibility of a parent-to-child nasal microbiome transplant. The investigators will test parent-to-neonate nasal microbiome transplantation as an intervention to reduce S. aureus acquisition in neonates. Neonates admitted to the Johns Hopkins Hospital neonatal intensive care unit (NICU) will be screened and parents will be approached for enrollment in the study. After consent and baseline screening of parents and neonates, eligible neonates will undergo a nasal microbiome transplant. This pilot study looks to determine whether transferring a parents healthy, diverse nasal microbiota to the infant(s) will create a healthy, diverse neonatal nasal microbiome. The investigators are planning an upcoming randomized controlled trial of this intervention and hope to establish feasibility during this pilot study.

ELIGIBILITY:
Inclusion Criteria:

Neonate:

1. Neonate has anticipated NICU length of stay > 7 days
2. Neonate ≥25 weeks gestation
3. At least one parent/adult provider not colonized with S. aureus (as determined by baseline screening)
4. Neonate is not colonized with S. aureus on baseline screening

Parent/adult provider:

1. Parent/adult provider is able to provide informed consent.

Exclusion Criteria:

Neonate:

1. Neonate has had a prior clinical or surveillance culture grow S. aureus
2. Neonate is a ward of the State
3. Neonate with antenatal suspicion for immunodeficiency (e.g. sibling with known immunodeficiency, genetic syndrome with known associated immunodeficiency)
4. Neonate cannot have nasal swabs collected (due to anatomic or other clinical intervention, including nasal packing)

Parent/adult Provider:

1. Parent/adult provider had positive COVID-19 test in prior 21 days
2. Parent/adult provider with signs or symptoms of respiratory illness (e.g. runny nose, congestion, fever, cough)
3. Parent/adult provider has been in close contact with someone in the last 7 days who had a respiratory viral infection, like the cold or the flu?
4. Parent/adult provider tests positive on baseline screening test for S. aureus nasal colonization.
5. Parent/adult provider tests positive on baseline screening test for a respiratory pathogen.
6. Parent/adult provider is not able to provide written informed consent
7. Parent/adult provider is not able to be present at the bedside at the time of intervention.
8. Parent/adult provider has history of chronic sinusitis, cystic fibrosis, or an infection with a multi-drug resistant organism.
9. Inability or unwillingness to complete the Donor questionnaire or a positive response to any question on the Donor questionnaire

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal nasal microbiome diversity after intervention | Day 4, 7, 10, 14 days post-intervention
  This outcome will be determined by analysis of periodic surveillance swabs collected after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Milstone, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States